CLINICAL TRIAL: NCT01556100
Title: Long-Term Vesicular Monoamine Transporter II Imaging and Clinical Assessment of Parkinson's Disease Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 99-3989A
Record Dates: First submitted 2012-03-06; First posted 2012-03-16 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2016-11

CONDITIONS: Parkinson Disease
Keywords: 18F-DTBZ AV-133 imaging
MeSH Terms: conditions — Parkinson Disease | interventions — florbenazine F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DTBZ AV-133 (Experimental): 18F-DTBZ AV-133 imaging
  Interventions: Drug: 18F-DTBZ AV-133

INTERVENTIONS:
Drug: 18F-DTBZ AV-133 — A total 40 PD subjects will be included in this study. PD subjects between 20 and 80 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, and blood test.

SUMMARY:
A total 40 PD subjects will be included in this study. PD subjects between 20 and 80 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, and blood test.

DETAILED DESCRIPTION:
The primary objective of this protocol is to assess the rate of change in striatal 18F-DTBZ uptake in a cohort of Parkinson's disease patients.

This study is expected to be completed in a period of 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 20 years to 80 years.
2. Patients should be fulfilled Criteria of diagnosis of Parkinson disease of "possible" or "probable" PD1.
3. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent)

Exclusion criteria:

1. Significant recent (within 6 months) history of neurological (including stroke and brain trauma) or psychiatric disorder.
2. Alcohol or substance abuse.
3. History or presence of QTc prolongation. (>500msec)
4. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
5. Unable to stay still in the MRI or PET scanner for 30 minutes.
6. Pregnancy and breast feeding.
7. Hepatic dysfunction with liver function test (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) of > 3x the upper limit of normal

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 18F-DTBZ AV-133
Started | 40
Completed | 34
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | 18F-DTBZ AV-133
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 55.08 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Region of Enrollment [Number; unit: participants]
  Taiwan | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in 18F-DTBZ Uptake in a Cohort of Parkinson's Disease Patients From Baseline to Month 36
Description: To expand the database of 18F-DTBZ PET imaging in Parkinson's Disease patients to refine the definition of a positive scan in patient with PD.
Time Frame: three years
Measure: Mean (80% Confidence Interval); unit: SUVR
Arm/Group | 18F-DTBZ AV-133
Number analyzed (Participants) | 34
SUVR | 12.95 [1.74 to 24.16]

2. Secondary Outcome: To Determine the Test/Retest 18F-DTBZ PET Measurements of Vesicular Monoamine Transporter II Binding in PD Patients.
Description: The test/retest reliability will be estimated from a subgroup of the study subjects (10 subjects) who receive additional scan within 4 weeks since baseline image.
  In order to refine the definition of a positive 18F-DTBZ in patient with PD as compared to healthy control, quantitative measurement will be used. The standard uptake value (SUV) of each brain regions will be calculated. The SUV is a widely used, simple PET quantifier, calculated as a ratio of tissue radioactivity concentration (e.g. in units kBq/ml) at time t, CPET(t) and injected dose (e.g. in units MBq) at the time of injection divided by body weight (e.g. in units kg).SUV = CPET(t) / (Injected dose / Patient's weight), t =90min, and the unit of SUV is g/ml.
Time Frame: three years
Population: A subgroup of 10 subjects receive additional scan for a test/retest reliability study
Measure: Mean (80% Confidence Interval); unit: g/mL
Arm/Group | 18F-DTBZ AV-133
Number analyzed (Participants) | 10
g/mL | 12.95 [1.74 to 24.16]

ADVERSE EVENTS:
Time Frame: three yaers
Arm/Group | 18F-DTBZ AV-133
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No